CLINICAL TRIAL: NCT02289001
Title: Study to Evaluate the Use of the SBAR (Situation-Background-Assessment-Recommendation) Checklist as a Means to Help Undergraduate Nursing Students Understand Team Member Roles and Improve Healthcare Team Communication
Brief Title: Simulation Training in Undergraduate Nursing Education as a Means to Improve Awareness of Team Member Roles
Acronym: SBAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Girona (Other)
Responsible Party: Principal Investigator, Marta Raurell-Torredà, Dr. Marta Raurell, Universitat de Girona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: SBAR-1
Record Dates: First submitted 2014-11-04; First posted 2014-11-13 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Communication
Keywords: patient simulation; simulation; teamwork; interdisciplinary health team; healthcare team; nursing; training programs
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education on SBAR worksheet (Experimental): Training in the use of the SBAR worksheet created to structure information exchange between healthcare professionals
  Interventions: Behavioral: Education on SBAR worksheet
- No education on SBAR worksheet (No Intervention): The control group will participate in the simulation without any prior training in teamwork skills beyond those included in the undergraduate nursing degree curriculum, which the intervention group also received.

INTERVENTIONS:
Behavioral: Education on SBAR worksheet — The intervention group will receive one hour of training in teamwork skills, distribution of roles and use of the SBAR worksheet before participating in the simulated scenario using a human patient simulator (HPS).
  Arms: Education on SBAR worksheet

SUMMARY:
Based on investigator's hypothesis, that incorporating the SBAR worksheet into the training of undergraduate Nursing students will increase their capacity to work in an interdisciplinary team, the investigators will assess whether introducing the SBAR improves the students' knowledge of their own role and that of others on the team (medical students), strengthens communication between team members, and enhances the quality of the patient assessment and interventions demonstrated by the nursing students caring for a critical patient (represented by a high-fidelity mannequin, a Human Patient Simulator).

DETAILED DESCRIPTION:
Students assigned to the intervention group will receive one hour of additional training in teamwork skills, communication between team members, and the relationship with patient safety, as well as how to distribute roles and responsibilities and how to use the SBAR worksheet. They will not be given the materials used to present the training session (PowerPoint slides, videos, and the SBAR worksheet) in order to avoid their sharing this information directly with students in the control group.

Training provided the Intervention Group

1. Basic competencies of healthcare professionals (Institute of Medicine, IOM, 2003) and of working as a team member (Interprofessional Education Collaborative (IPEC). Core competencies for Interprofessional Collaborative Practice. 2011. Available at: http://www.aacn.nche.edu/education-resources/ipecreport.pdf)
2. Use of the SBAR (Situation-Background-Assessment-Recommendation) worksheet in accordance with the Kaiser Permanente Guidelines for Communicating with Physicians Using the SBAR Process. Available at: http://fliptheclinic.org/wordpress/wp-content/uploads/community_uploads/1598/SBAR%20Guidelines%20Kaiser%20Permanente.pdf. Accessed Oct 17, 2014):
3. Distribution of roles and responsibilities of the interdisciplinary care team for a critical patient (airway management, assessment nurse/physician, medication nurse, procedure nurse, documenting nurse)

On a day when clinical practice is scheduled, according to the 2014-2015 academic year, the students will report to the simulation laboratory. All students in both study arms will participate in a simulated scenario, with cases validated by the National League for Nursing, in a setting that mimics an emergency department with a critical patient (HPS) in a state of shock. Three nursing students and a medical student will intervene in each scenario. If the scenario requires an additional intervention to guide the students or redirect situations that reach an impasse, a professor will be prepared to take on the role of an emergency room physician or nursing supervisor.

Students who do not receive the complementary training (i.e., the control group) will be directed to a different laboratory than the intervention group while they wait to be called for their participation in the simulated scenario.

Ten minutes before beginning the scenario, each group (control and intervention) will receive the documents corresponding to the simulated patient's clinical history. Students in the intervention group will also have a printed SBAR worksheet, which they will be familiar with because of the complementary training. This worksheet will be mixed with the documents related to the patient's clinical history so that the professors participating in the scenario and those doing the evaluation will not be readily able to identify which study arm in participating in a given scenario.

A professor will randomize the scenarios, following the codes delivered in sealed envelopes and that were previously assigned a number directly linked to the corresponding study arm (intervention, control). The envelopes will be kept in a locked box in the simulation laboratory, and will be opened each day of clinical practice by a professor not involved in the study.

Sample size To calculate the necessary sample, we considered the difference in medians observed in a previous study in the same population (Raurell-Torredà M, Olivet-Pujol J, Romero-Collado A, Malagon-Aguilera MC, Patiño-Masó, J, Baltasar-Bagué A. Case-based learning and simulation: useful tools to enhance nurses' education? Non-randomized controlled trial". J Nurs Scholarsh. 2014, Oct 25. doi: 10.1111/jnu.12113). The standardized median difference was 0.9 points. With the aim of obtaining the same difference in the present study, accepting an alpha risk of 0.05 and beta risk less than 20% in a two-tailed test, the estimated sample size 21 scenarios in each arm of the study.

Statistical analysis Qualitative variables will be expressed as frequency and percentage, using the Chi square or Fisher test to compare groups, as appropriate. Quantitative variables will be shown mean and standard deviation (SD) or median and interquartile range (P25-P75), depending on the normality of the distribution, and groups will be compared using Student t or Mann-Whitney U test, respectively. A P-value <0.05 will be considered significant. All analyses will be done using IBM SPSS Statistics (IBM Statistics®, Markham, ON, Canada).

Given the impossibility of predicting how students who do not participate in the simulation would have behaved, losses to follow-up will be managed per protocol rather than intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Passing grade on the emergency care topics in the required course "Adult Patient II", which focuses on nursing care planning related to various clinical pathologies or syndromes and surgical procedures
* Current student in the required course "Techniques and Procedures III", which incorporates simulation related to Clinical Nursing II and Psychology course content

Exclusion criteria:

- No signed informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the use of the SBAR checklist as a means to help undergraduate nursing students identify their own role, understand the roles of other health professionals (assess skill level (KidSIM Team Performance Scale) | During the 2-month data collection period, changes in skill level will be measured during the simulation scenario for each study arm, using an assessment scale (KidSIM Team Performance Scale) validated for this purpose.
  The study will use the KidSIM Team Performance Scale, designed and validated by Sigalet et al. for use in undergraduate nursing, medicine and physiotherapy degree programs. The KidSIM scale has 5 items about roles and 6 about communication.

SECONDARY OUTCOMES:
Evaluation of the SBAR instrument to improve patient assessment and intervention skills of undergraduate nursing students using human patient simulators (assess skill level using the Wolf scale) | During the 2-month data collection period, changes in skill level will be measured during the simulation scenario for each study arm, using an assessment scale (Wolf) validated for this purpose).
  The Wolf scale was specifically designed to evaluate nontechnical skills (critical thinking and patient safety, communication, assessment, diagnosis and intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Marta Raurell, RN, PhD, Principal Investigator — Universitat de Girona

REFERENCES:
- [Background] Sigalet E, Donnon T, Cheng A, Cooke S, Robinson T, Bissett W, Grant V. Development of a team performance scale to assess undergraduate health professionals. Acad Med. 2013 Jul;88(7):989-96. doi: 10.1097/ACM.0b013e318294fd45. PMID 23702524
- [Background] Henneman EA, Cunningham H, Roche JP, Curnin ME. Human patient simulation: teaching students to provide safe care. Nurse Educ. 2007 Sep-Oct;32(5):212-7. doi: 10.1097/01.NNE.0000289379.83512.fc. PMID 17828022
- [Background] Raurell-Torreda M, Olivet-Pujol J, Romero-Collado A, Malagon-Aguilera MC, Patino-Maso J, Baltasar-Bague A. Case-based learning and simulation: useful tools to enhance nurses' education? Nonrandomized controlled trial. J Nurs Scholarsh. 2015 Jan;47(1):34-42. doi: 10.1111/jnu.12113. Epub 2014 Oct 25. PMID 25346329
- [Background] Wolf L, Dion K, Lamoureaux E, Kenny C, Curnin M, Hogan MA, Roche J, Cunningham H. Using simulated clinical scenarios to evaluate student performance. Nurse Educ. 2011 May-Jun;36(3):128-34. doi: 10.1097/NNE.0b013e318216120b. PMID 21502849